CLINICAL TRIAL: NCT00321646
Title: A Phase II Study of Neoadjuvant Bevacizumab Plus Docetaxel in High Risk Patients With Prostate Cancer Undergoing Radical Prostatectomy
Brief Title: Neoadjuvant Bevacizumab Plus Docetaxel in High Risk Patients With Prostate Cancer Undergoing Radical Prostatectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mary-Ellen Taplin, MD (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Duke University (Other); Genentech, Inc. (Industry); Sanofi (Industry)
Responsible Party: Sponsor-Investigator, Mary-Ellen Taplin, MD, Assistant Professor of Medicine, HMS, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-438
Record Dates: First submitted 2006-05-02; First posted 2006-05-04 (Estimated); Results first posted 2013-12-25 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-04

CONDITIONS: Prostate Cancer; Adenocarcinoma of the Prostate
Keywords: prostate cancer; bevacizumab; docetaxel; radical prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Bevacizumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- chemotherapy (Experimental): docetaxel and bevacizumab prior to prostatectomy
  Interventions: Drug: Bevacizumab; Drug: Docetaxel

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab (marketed as Avastin, Genentech) is an antibody to all isoforms of vascular endothelial growth factor and is the first putative anti-angiogenic agent approved by the Food and Drug Administration (FDA) for the treatment of cancer.All subjects will be treated with intravenous docetaxel and bevacizumab for 5 cycles, followed by docetaxel alone for Cycle 6. Bevacizumab will be given first, at a starting dose of 15 mg/kg. Bevacizumab will be given once every 21 days in the infusion center.
  Other Names: Avastin
Drug: Docetaxel — Docetaxel will be given intravenously once every 21 days in the infusion center. The starting dose is 70mg/square meter.
  Other Names: Taxotere

SUMMARY:
The main purpose of this trial is to collect information and to evaluate the effects, good or bad, the combination of docetaxel and bevacizumab has on patients with high risk prostate cancer that are undergoing radical prostatectomy.

DETAILED DESCRIPTION:
* Patients who are eligible for this study will undergo an endorectal MRI scan test before beginning the research study.
* After the MRI, the patient will begin the docetaxel plus bevacizumab part of the study. Each treatment cycle starts on the day you receive both drugs and lasts 21 days. Patients will undergo a total of 6 cycles-5 with docetaxel plus bevacizumab and one with docetaxel alone.
* At the beginning of each cycle, the patient will come into the clinic for a visit that will last about 3 hours. The following will happen at these visits: physical examination including vital signs and rectal exam; questions about the patients health and the medications they are taking; blood tests (both routine and research blood tests); urine tests; bevacizumab infusion; docetaxel infusion.
* The patients first dose of bevacizumab will be given on Day 1 of the first cycle over 90 minutes. If the patient tolerates the 90-minute infusion well, later doses may be given over a shorter period of time.
* The day before and the morning of the beginning of each cycle, the patient will be given a steroid called dexamethasone in pill form to help decrease the side effects of the treatment.
* The above tests and procedures will be repeated every 21 days a total of five times. For the sixth time, the patient will have all the same tests and procedures except they will not receive bevacizumab.
* After the six cycles, the patient will undergo another endorectal MRI.
* One to two months after finishing the sixth cycle, the patient will undergo a radical prostatectomy to remove their prostate.
* Two to three months after the surgery the patient will return to the clinic to have the following tests and procedures: questions about the patient's health; routine blood tests and research blood tests.

ELIGIBILITY:
Inclusion Criteria:

* Histological documentation of adenocarcinoma of the prostate, with available biopsy pathology. Material from this biopsy must be available for central review at DF/HCC by the beginning of the second cycle of therapy.
* Potential candidate for radical prostatectomy
* Must meet one or more of the below characteristics: Gleason score of 8, 9 or 10; serum PSA of greater than or equal to 20 ng/mL; clinical T stage of T3; PSA velocity of greater than or equal to 2ng/mL/year in the year prior to diagnosis; Gleason score of 7 and erMRI T3 disease; Greater than or equal to 50% of the total number of biopsy cores positive for prostate cancer and either PSA > 10ng/mL or Gleason score of 7 or clinical T stage of T2a, T2b or T2c.
* Greater than six weeks since any major surgery
* Serum testosterone > 100ng/dL
* ECOG Performance Status of 0 or 1
* ANC > 1,500/ul
* Platelets > 100,000/ul
* Total bilirubin, alkaline phosphatase, AST and ALT within normal limits
* Creatinine < 2.0 x upper limit of normal

Exclusion Criteria:

* History of prior radiation, surgery or hormonal therapy treatment for prostate cancer
* Clinical evidence of metastatic prostate cancer
* Ongoing oral steroid use
* Pre-existing neuropathy of grade 2 or greater
* Severe claustrophobia, inability to lie still in a magnet for 60 minutes, a pacemaker, or any other condition that would preclude proximity to a strong magnet.
* History of the following conditions: unstable angina; symptomatic, clinically significant peripheral vascular disease; NY Heart Association Grade 2 or greater heart failure; uncontrolled hypertension; myocardial infarction or stroke < 12 months prior to enrollment; uncontrolled hypertension; active, uncontrolled infection; history of DVT, PE or known coagulopathy or bleeding diathesis; ongoing us of anticoagulant therapy; history of abdominal fistulas, GI perforation, or intra-abdominal abscess within 6 months prior to study entry; non-healing ulcer or fracture; history of another malignancy diagnosed within the last five years; spot urine protein: creatinine ratio > 1.0 at screening.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2006-06; Primary Completion 2008-11 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary-Ellen Taplin, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- [Derived] Karlou M, Tzelepi V, Efstathiou E. Therapeutic targeting of the prostate cancer microenvironment. Nat Rev Urol. 2010 Sep;7(9):494-509. doi: 10.1038/nrurol.2010.134. PMID 20818327

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 42 subjects were consented, screened, registered and enrolled between 7/27/06 and 3/24/09 in the relevant clinics at Duke University (5 subjects) and DF/HCC (37 subjects).
Pre-assignment Details: No subjects were found to be ineligible after signing the informed consent form and registering with the QACT.
Groups:
- Chemotherapy: docetaxel and bevacizumab prior to prostatectomy
  Docetaxel : Docetaxel will be given intravenously once every 21 days in the infusion center. The starting dose is 70mg/square meter.
  Bevacizumab : Bevacizumab (marketed as Avastin, Genentech) is an antibody to all isoforms of vascular endothelial growth factor and is the first putative anti-angiogenic agent approved by the Food and Drug Administration (FDA) for the treatment of cancer.All subjects will be treated with intravenous docetaxel and bevacizumab for 5 cycles, followed by docetaxel alone for Cycle 6. Bevacizumab will be given first, at a starting dose of 15 mg/kg. Bevacizumab will be given once every 21 days in the infusion center.
Period: Neoadjuvant Chemotherapy
Arm/Group | Chemotherapy
Started | 42
Completed | 38 (1 pt withdrew before start of therapy, 38 completed 6 cycles neoadjuvant therapy.)
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 2
Not completed — Disease progression | 1
Period: Prostatectomy
Arm/Group | Chemotherapy
Started | 37
Completed | 37
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 42 enrolled, 1 participant withdrew before receiving treatment.
Arm/Group | Chemotherapy
Number analyzed (Participants) | 41
Age, Continuous [Median (Full Range); unit: year]
  Between 18 and 65 years | 55 [41 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 41
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Endorectal MRI Response After Completion of 6 Cycles of Neoadjuvant Therapy
Description: A response was defined as a decrease in tumor size of >50% for the largest lesion in the prostate by endorectal MRI.
Time Frame: after 6 months of neoadjuvant chemotherapy.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Chemotherapy
Number analyzed (Participants) | 41
proportion of participants | 0.29 [0.16 to 0.45]

2. Secondary Outcome: PSA Response After Completing 6 Cycles of Neoadjuvant Chemotherapy.
Description: The rate of PSA decline by 50% compared to baseline PSA.
Time Frame: after 6 months of ajuvant chemotherapy.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Chemotherapy
Number analyzed (Participants) | 41
proportion of participants | 0.22 [0.11 to 0.38]

ADVERSE EVENTS:
Time Frame: 6 months during the neoadjuvant chemotherapy.
Arm/Group | Chemotherapy
Serious Adverse Events (participants affected / at risk) | 11/41
Other Adverse Events (participants affected / at risk) | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy (N=41)
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Allergic reaction (Immune system disorders) | 1
Infection w/ unk ANC skin (cellulitis) (Infections and infestations) | 1
Leukocytes (Investigations) | 1
Lymphopenia (Investigations) | 3
Neutrophils (Investigations) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy (N=41)
Hyperglycemia (Metabolism and nutrition disorders) | 37
Fatigue (General disorders) | 33
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 22
Alopecia (Skin and subcutaneous tissue disorders) | 19
Taste disturbance (Nervous system disorders) | 17
Insomnia (Psychiatric disorders) | 16
Tearing (Eye disorders) | 15
Nausea (Gastrointestinal disorders) | 15
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 12
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 12
Hemoglobin (Blood and lymphatic system disorders) | 11
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 11
Nail changes (Skin and subcutaneous tissue disorders) | 11
Bicarbonate (Metabolism and nutrition disorders) | 10
Neuropathy-sensory (Nervous system disorders) | 10
Head/headache (Nervous system disorders) | 9
Constipation (Gastrointestinal disorders) | 8
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 8
AST, SGOT (Investigations) | 8
Anorexia (Metabolism and nutrition disorders) | 8
Vision-blurred (Eye disorders) | 7
Joint, pain (Musculoskeletal and connective tissue disorders) | 7
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 7
Dyspepsia (Gastrointestinal disorders) | 6
Fever w/o neutropenia (General disorders) | 6
Allergic reaction (Immune system disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Hypertension (Vascular disorders) | 5
Lymphopenia (Investigations) | 4
Hyponatremia (Metabolism and nutrition disorders) | 4
Anxiety (Psychiatric disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 4
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 4
Sweating (Skin and subcutaneous tissue disorders) | 4
Ocular-other (Eye disorders) | 3
Flatulence (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Rigors/chills (General disorders) | 3
Edema limb (General disorders) | 3
Pain NOS (General disorders) | 3
Pain-other (General disorders) | 3
ALT, SGPT (Investigations) | 3
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 3
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 3
Depression (Psychiatric disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No